CLINICAL TRIAL: NCT01316783
Title: Genetics of Obesity, Diabetes, and Heart Disease in African Diaspora Populations
Status: Enrolling by invitation | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110110; 11-HG-0110
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-22

CONDITIONS: Diabetes; Cardiovascular Disease
Keywords: Cardiometabolic Diseases; Natural History
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: African ancestry and whites (who will serve as a comparison group)

SUMMARY:
Background:

- African Americans have one of the highest rates of type 2 diabetes in the United States, and often have other medical problems related to obesity and cardiovascular disease. These conditions have various risk factors, including high blood sugar levels, high cholesterol levels, and insulin resistance. However, these risk factors have not been studied very closely in individuals with African ancestry, including Afro-Caribbean and sub-Saharan Africa migrant populations. Researchers are interested in conducting a genetic study on obesity, adult-onset diabetes, heart disease, and other common health conditions in individuals with African ancestry.

Objectives:

- To collect genetic and non-genetic information from individuals with African ancestry to study common health conditions related to obesity, adult-onset diabetes, and heart disease.

Eligibility:

- Individuals at least 18 years of age who self-identify as African American, Afro-Caribbean, or migrants from sub Saharan Africa.

Design:

* Participants will undergo a physical examination and will provide a blood sample for study.
* Participants will also answer questions about personal and family medical history and current lifestyle behaviors.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
Study Design:

The study is comprised of a population-based sample from Dr. Anne Sumner s ongoing NIDDK studies to perform a quantitative trait analysis of multiple metabolic biomarkers and disorders including T2D, hypertension, CVD and obesity in a total of 1000 people of African ancestry and approximately100 whites (who will serve as a comparison group) residing in the United States. Because some of the identified variants will be rare, we will use the methods proposed by Li and Leal. Under an additive model and at a MAF of 0.04, this sample size has 80% power to detect a genetic effect that may explain a 1-4 unit change depending on the trait in question (e.g., BMI in kg/m^2, blood glucose in mg/dL, systolic and diastolic BP in mmHG).

We will also perform exome sequencing of 48 cases of African descent and genotype identified variants in the larger cohort. Cases for exome sequencing will consist of individuals who have more than one metabolic condition, i.e., diabetes, pre-diabetes, obesity, hypertension and/or dyslipidemia. We propose to carry out exome capture of 48 individuals (96 chromosomes). Given the probability of observing a specific allele one or more times of 1 - (1-p)^2N (where p is the minor allele frequency), a sample of 48 individuals (96 chromosomes) provides a 99% probability of finding a sequence variant with a minor allele frequency (MAF) of 0.05, 98% probability of finding a variant with an MAF of 0.04, 95% probability of finding a variant with an MAF of 0.03, 86% probability of finding a variant with an MAF of 0.02 and 62% probability of finding a variant with an MAF of 0.01. We will use four main filters to identify potential variants with functional consequences. We will look for 1) SNPs that are intragenic or in promoter regions, 2) SNPs that cause nonsynonymous coding changes, 3) nonsense mutations, and 4) missense mutations that have possible or probable damaging protein effects. All selected SNPs will be tested for potential association with all metabolic parameters in this study.

Primary Objective:

Genotype variants of interest from genetic epidemiology studies conducted in Dr. Rotimi s lab in these individuals, with thorough clinical measurements available, in order to investigate biological mechanisms underlying observed associations.

Secondary Objectives:

Conduct whole-exome capture on a subset of cases with at least 2 metabolic disorders (i.e., diabetes, pre-diabetes, obesity, hypertension and/or dyslipidemia). Genotype identified variants in the larger cohort of 1000 persons or in existing studies of African ancestry individuals (Howard University Family Study or Africa America Diabetes Mellitus Study).

Exploratory Objectives:

Endpoints: Obesity, Metabolic Syndrome, Dyslipidemia, Pre-Diabetes, and Diabetes

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will include unrelated persons who self-identify as white or African American, Afro-Caribbean or migrant from sub-Saharan Africa. Adults of African ancestry are prioritized for this study because of the paucity of genetics studies investigating the association of risk alleles contributing to the prevalence of T2D, CVD, obesity and other common conditions in this population. A small proportion of whites (less than 10%) will be included in this study, as they are in Dr. Sumner s ongoing projects; they will have the same clinical measurements obtained in the same laboratory to serve as a comparison group. This study only includes adults because these phenotypes are more commonly present in adults. In summary, inclusion criteria include:

* Persons who self-identify as either

  * African American
  * Afro-Caribbean
  * A migrant from sub-Saharan Africa
  * White
* Persons >= 18 years
* Participation in a protocol with Dr. Anne Sumner, NIDDK/NIH

EXCLUSION CRITERIA:

Related individuals are excluded to avoid biases in our analyses due to genomic similarities between people who are related. No prisoners will be included in this study. Pregnant women are excluded from this study because pregnancy induces changes in metabolism that would interfere with the measurements and outcomes of the study. In summary, exclusion criteria include:

* Individuals related to participants
* Prisoners
* Pregnant women

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The estimated number of participants is 1100 with 100 of those being white participants. Based on Dr. Sumner's previous work with these cohorts, we expect 25% of the African Ancestry populations to have abnormal glucose tolerance or diabetes, 50 percent to be obese, and 20% to be hypertensive. For whites the % frequency will be lower. The power analysis is based on black populations, the focus of the study. The enrollment ceiling is 1100 and the anticipated enrollment by year is 100 individuals.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2011-05-06 (Actual)

PRIMARY OUTCOMES:
Metabolic disorders | One study visit
  type 2 diabetes, metabolic outcomes, dyslipidemia

CONTACTS AND LOCATIONS:
Overall Officials: Charles N Rotimi, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared through dbGAP following completion of data collection and planned assays.
Supporting Information: Study Protocol
Time Frame: Within 3 months after the last data generated.
Access Criteria: Data will be shared through dbGaP with controlled access based on IRB approval: requestor must provide documentation of local IRB approval.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-HG-0110.html